CLINICAL TRIAL: NCT07325851
Title: Prospective and Observational Study of Patients Referred to the Chronic Pain Unit for Palliative Treatment With Ozone Therapy Between 2026 and 2029. Prospective Study EPOOzo-2.
Brief Title: Patients Referred to the Chronic Pain Unit for Palliative Treatment With Ozone Therapy Between 2026 and 2029.
Acronym: EPOOzo-2
Status: Not yet recruiting | Type: Observational
Sponsor: Bernardino Clavo, MD, PhD (Other)
Collaborators: Dr. Negrin University Hospital (Other); Fundacion Canaria Instituto de Investigacion Sanitaria de Canarias (Other); Complejo Hospitalario Universitario Insular Materno Infantil (CHUIMI) (Unknown); Instituto Universitario de Microelectrónica Aplicada de la Universidad de Las Palmas de Gran Canaria (IUMA-ULPGC) (Unknown); Council of Gran Canaria (Other)
Responsible Party: Sponsor-Investigator, Bernardino Clavo, MD, PhD, Principal Investigator, Research Unit Director, Dr. Negrin University Hospital
Organization: Dr. Negrin University Hospital (Other)
Other Study IDs: 2025-642-1; 0177-2025-OBS (Registry Identifier: Identificador REEC)
Record Dates: First submitted 2025-12-23; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Chemotherapy-Induced Peripheral Neuropathy; Radiation Toxicity; Chronic Pain; Delayed Wound Healing; Refractory Symptoms
Keywords: Ozone Therapy; Health-related quality of life; Chemotherapy-induced Peripheral Neuropathy; Radiation-induced toxicity; Hyperspectral imaging; Infrared imaging; Heart Rate Variability; Sudoscan; Vibrometry; Oxidative stress; Gut Microbiota; Anxiety and Depression
MeSH Terms: conditions — Radiation Injuries; Chronic Pain; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 40 Weeks
Biospecimen Retention: Samples With DNA — Blood and stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ozone Group: Patients with refractory symptoms referred for palliative treatment with ozone therapy between 2026 and 2029.
  Interventions: Procedure: Ozone Therapy

INTERVENTIONS:
Procedure: Ozone Therapy — Systemic (rectal, autohemotherapy) and/or local ozone administration (cutaneous, intravaginal, intravesical). Dosage, frequency, and duration will depend on the symptoms treated and clinical evolution. Usually planned 40 sessions over 4 months.
  Other Names: Ozone Treatment

SUMMARY:
The main objective of this study is to analyze the impact on the health-related quality of life of patients with refractory symptoms who have been referred to the Dr. Negrín University Hospital Chronic Pain Unit for adjuvant palliative treatment with ozone therapy between January 2026 and December 2029. Additionally, the study aims to evaluate several specific symptoms, hyperspectral and thermal images, non-invasive clinical parameters related to the Autonomic Nervous System (such as heart rate variability, electrochemical skin conductance, and vibration perception thresholds), oxidative stress and inflammatory parameters, and gut microbiota composition.

DETAILED DESCRIPTION:
Patients are referred to the Chronic Pain Unit in the absence or failure of standard treatment, or when the standard treatment is associated with high morbidity or high risk. Frequently, these patients present alterations in self-perceived health-related quality of life (HRQoL), anxiety, depression, and other symptoms such as radiation-induced pelvic toxicity or chemotherapy-induced peripheral neuropathy (CIPN).

This prospective observational study (EPOOzo-2) aims to evaluate the effect of adjuvant symptomatic/palliative ozone therapy on HRQoL and potential changes from baseline. Specifically, it incorporates new non-invasive technologies to objectively assess microcirculation, neuropathy and autonomic regulation.

Main Objectives:

1. Analyze the impact on HRQoL of patients with refractory symptoms treated with ozone.

Secondary Objectives: Depending on the clinical case, analyze the impact of ozone treatment on: 2. Anxiety and depression. 3. Treated symptoms (e.g., pain, paresthesia). 4. Fatigue. 5. Toxicity grade (in cancer patients). 6. Non-invasive clinical parameters related to the Autonomic Nervous System (central and peripheral) and somatosensory function. 7. Biochemical parameters and gut microbiome analysis (in patients with systemic/rectal ozone).

Methodology: Prospective and observational study of patients referred for symptomatic/palliative ozone therapy between January 2026 and December 2029.

Assessments at weeks: 0 (baseline), 16 (end of O3/O2 treatment), 28 (12 weeks after the end of ozone), and 40 (24 weeks after the end of ozone).

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults ≥ 18 years old.
* 2. Patients referred to the Chronic Pain Unit of the Dr. Negrín University Hospital for symptomatic/palliative treatment with ozone therapy because conventional treatment does not exist, has failed, has offered insufficient results, or is associated with high risk/morbidity.
* 3. After evaluation of symptoms and patients, it exists a potential benefit of adding ozone treatment to the current treatment.
* 4. Patients have no contraindications for ozone treatment.
* 5. Patients must sign the specific Informed Consent for this study and for the ozone treatment.

Exclusion Criteria:

* 1. Age < 18 years old.
* 2. Psychiatric illness or social situations that would limit compliance with study requirements.

Contraindication or disability to attend scheduled treatments.

* 3. Contraindication or disability to attend scheduled treatments.
* 4. Uncontrolled clinical conditions (e.g., severe heart failure, massive hemorrhage, status epilepticus).
* 5. Life expectancy < 6 months.
* 6. Known allergy to ozone.
* 7. Hemochromatosis (for systemic ozone treatment).
* 8. Pregnancy (for systemic ozone treatment).
* 9. Significant Glucose-6-Phosphate Dehydrogenase deficiency (Favism) (for systemic ozone treatment).
* 10. Patients who do not meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients submitted to the Chronic Pain Unit of the Hospital Universitario de Gran Canaria Dr. Negrín, between January 2026 and December 2029, for symptomatic/palliative treatment with ozone therapy because standard treatment does not exist, it has been unsuccessful, or it is associated with high risk or high morbidity.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-01-14 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Health-Related Quality of Life by the "EQ-5D-5L" Questionnaire (at the end of ozone therapy). | At the end of ozone therapy (approx. week 16).
  Self-reported evaluation of 5 physical and emotional items scored in five levels, plus a Visual Analog Scale (EQ-VAS) from 0 (worst health) to 100 (best health).

SECONDARY OUTCOMES:
Change from Baseline in Health-Related Quality of Life by the "EQ-5D-5L" Questionnaire (at 12 weeks after the end of ozone therapy). | At 12 weeks after the end of ozone therapy (approx. week 28).
  Self-reported evaluation of 5 physical and emotional items scored in five levels, plus a Visual Analog Scale (EQ-VAS) from 0 (worst health) to 100 (best health).
Change from Baseline in Health-Related Quality of Life by the "EQ-5D-5L" Questionnaire (at 24 weeks after the end of ozone therapy). | At 24 weeks after the end of ozone therapy (approx. week 40).
  Self-reported evaluation of 5 physical and emotional items scored in five levels, plus a Visual Analog Scale (EQ-VAS) from 0 (worst health) to 100 (best health).
Change from Baseline in Anxiety and Depression Levels (HAD Scale) (at the end of ozone therapy). | At the end of ozone therapy (approx. week 16).
  Hospital Anxiety and Depression Scale (HADS). Scores range from 0 to 21 for each subscale, where higher scores indicate worse anxiety or depression.
Change from Baseline in Anxiety and Depression Levels (HAD Scale) (at 12 weeks after the end of ozone therapy). | At 12 week after the end of ozone therapy (approx. week 28).
  Hospital Anxiety and Depression Scale (HADS). Scores range from 0 to 21 for each subscale, where higher scores indicate worse anxiety or depression.
Change from Baseline in Anxiety and Depression Levels (HAD Scale) (at 24 weeks after the end of ozone therapy). | At 24 week after the end of ozone therapy (approx. week 40).
  Hospital Anxiety and Depression Scale (HADS). Scores range from 0 to 21 for each subscale, where higher scores indicate worse anxiety or depression.
Change from Baseline in Health-Related Quality of Life by the "QLQ-C30" Questionnaire (only in cancer patients). (At the end of ozone therapy). | At the end of ozone therapy (approx. week 16).
  The EORTC QLQ-C30 is a 30-item questionnaire that includes five functional scales (physical, role, emotional, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, and pain), a global health status scale, and several single items. Scores are transformed to a 0-100 scale. For functional and global health scales, higher scores represent better functioning or quality of life. For symptom scales/items, higher scores indicate greater symptomatology or problems
Change from Baseline in Health-Related Quality of Life by the "QLQ-C30" Questionnaire (only in cancer patients). (At 12 weeks after the end of ozone therapy). | At 12 weeks after the end of ozone therapy (approx. week 28).
  The EORTC QLQ-C30 is a 30-item questionnaire that includes five functional scales (physical, role, emotional, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, and pain), a global health status scale, and several single items. Scores are transformed to a 0-100 scale. For functional and global health scales, higher scores represent better functioning or quality of life. For symptom scales/items, higher scores indicate greater symptomatology or problems
Change from Baseline in Health-Related Quality of Life by the "QLQ-C30" Questionnaire (only in cancer patients). (At 24 weeks after the end of ozone therapy). | At 24 weeks after the end of ozone therapy (approx. week 40).
  The EORTC QLQ-C30 is a 30-item questionnaire that includes five functional scales (physical, role, emotional, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, and pain), a global health status scale, and several single items. Scores are transformed to a 0-100 scale. For functional and global health scales, higher scores represent better functioning or quality of life. For symptom scales/items, higher scores indicate greater symptomatology or problems
Change from Baseline in Fatigue (Chalder Fatigue Scale and/or EORTC QLQ-FA12 for cancer patients) (at the end of ozone therapy). | At the end of ozone therapy (approx. week 16).
  Assessed using the Chalder Fatigue Scale (CFQ-11) and/or EORTC QLQ-FA12 for cancer patients. Higher scores indicate greater fatigue
Change from Baseline in Fatigue (Chalder Fatigue Scale and/or EORTC QLQ-FA12 for cancer patients) (at 12 weeks after the end of ozone therapy). | At 12 weeks after the end of ozone therapy (approx. week 28).
  Assessed using the Chalder Fatigue Scale (CFQ-11) and/or EORTC QLQ-FA12 for cancer patients. Higher scores indicate greater fatigue
Change from Baseline in Fatigue (Chalder Fatigue Scale and/or EORTC QLQ-FA12 for cancer patients) (at 24 weeks after the end of ozone therapy). | At 24 weeks after the end of ozone therapy (approx. week 40).
  Assessed using the Chalder Fatigue Scale (CFQ-11) and/or EORTC QLQ-FA12 for cancer patients. Higher scores indicate greater fatigue
Change from Baseline in Pain Score (Visual Analog Scale), (at the end of ozone therapy). | At the end of ozone therapy (approx. week 16).
  Self-reported evaluation of pain severity using a Visual Analog Scale (VAS), scored from 0 ("No pain") to 10 ("Pain as bad as you can imagine").
Change from Baseline in Pain Score (Visual Analog Scale), (at 12 weeks after the end of ozone therapy). | At 12 weeks after the end of ozone therapy (approx. week 28).
  Self-reported evaluation of pain severity using a Visual Analog Scale (VAS), scored from 0 ("No pain") to 10 ("Pain as bad as you can imagine").
Change from Baseline in Pain Score (Visual Analog Scale), (at 24 weeks after the end of ozone therapy). | At 24 weeks after the end of ozone therapy (approx. week 40).
  Self-reported evaluation of pain severity using a Visual Analog Scale (VAS), scored from 0 ("No pain") to 10 ("Pain as bad as you can imagine").
Change from Baseline in the grade of toxicity secondary to cancer-treatment (if applicable) according to the CTCAE v5.0 scale, (at the end of ozone therapy). | At the end of ozone therapy (approx. week 16).
  Grade of toxicity secondary to cancer-treatment according to the CTCAE v5.0 (Common Terminology Criteria for Adverse Events from the National Cancer Institute) scale. Each toxicity is usually scored from 0 (asymptomatic or mild symptoms) to 5 (death).
Change from Baseline in the grade of toxicity secondary to cancer-treatment (if applicable) according to the CTCAE v5.0 scale, (at 12 weeks after the end of ozone therapy). | At 12 weeks after the end of ozone therapy (approx. week 28).
  Grade of toxicity secondary to cancer-treatment according to the CTCAE v5.0 (Common Terminology Criteria for Adverse Events from the National Cancer Institute) scale. Each toxicity is usually scored from 0 (asymptomatic or mild symptoms) to 5 (death).
Change from Baseline in the grade of toxicity secondary to cancer-treatment (if applicable) according to the CTCAE v5.0 scale, (at 24 weeks after the end of ozone therapy). | At 24 weeks after the end of ozone therapy (approx. week 40).
  Grade of toxicity secondary to cancer-treatment according to the CTCAE v5.0 (Common Terminology Criteria for Adverse Events from the National Cancer Institute) scale. Each toxicity is usually scored from 0 (asymptomatic or mild symptoms) to 5 (death).
Change from Baseline in Electrochemical Skin Conductance (Sudoscan), (at the end of ozone therapy). | At the end of ozone therapy (approx. week 16).
  Non-invasive evaluation of sudomotor function (small fiber neuropathy assessment). Measured in microsiemens (µS) on hands and feet using SUDOSCAN technology.
Change from Baseline in Electrochemical Skin Conductance (Sudoscan), (at 12 weeks after the end of ozone therapy). | At 12 weeks after the end of ozone therapy (approx. week 28).
  Non-invasive evaluation of sudomotor function (small fiber neuropathy assessment). Measured in microsiemens (µS) on hands and feet using SUDOSCAN technology.
Change from Baseline in Vibration Perception Thresholds (Multifrequency Vibrometry), (at the end of ozone therapy). | At the end of ozone therapy (approx. week 16).
  Assessment of large fiber nerve function using the VibroSense Meter II. Measures perception thresholds at different frequencies (e.g., 4Hz to 500Hz).
Change from Baseline in Vibration Perception Thresholds (Multifrequency Vibrometry), (at 12 weeks after the end of ozone therapy). | At 12 weeks after the end of ozone therapy (approx. week 28).
  Assessment of large fiber nerve function using the VibroSense Meter II. Measures perception thresholds at different frequencies (e.g., 4Hz to 500Hz).
Change from Baseline in Postural Stability (Equilibrium Platform), (at the end of ozone therapy). | At the end of ozone therapy (approx. week 16).
  Functional assessment of balance and Center of Pressure (CoP) displacement using specific force platforms.
Change from Baseline in Postural Stability (Equilibrium Platform), (at 12 weeks after the end of ozone therapy). | At 12 weeks after the end of ozone therapy (approx. week 28).
  Functional assessment of balance and Center of Pressure (CoP) displacement using specific force platforms.
Change from Baseline in Heart Rate Variability (HRV), (at the end of ozone therapy). | At the end of ozone therapy (approx. week 16).
  Non-invasive assessment of the Autonomic Nervous System (vagal tone) by analyzing time intervals between heartbeats (RR intervals).
Change from Baseline in Heart Rate Variability (HRV), (at 12 weeks after the end of ozone therapy). | At 12 weeks after the end of ozone therapy (approx. week 28).
  Non-invasive assessment of the Autonomic Nervous System (vagal tone) by analyzing time intervals between heartbeats (RR intervals).
Changes from baseline in Hyperspectral signatures and Infrared images obtained from hands and feet at the end of follow-up, (at the end of ozone therapy). | At the end of ozone therapy (approx. week 16).
  Assessment of the percentage of reflectance for each wavelength of the hyperspectral and infrared images obtained with specific devices.
Changes from baseline in Hyperspectral signatures and Infrared images obtained from hands and feet at the end of follow-up, (at 12 weeks after the end of ozone therapy). | At 12 weeks after the end of ozone therapy (approx. week 28).
  Assessment of the percentage of reflectance for each wavelength of the hyperspectral and infrared images obtained with specific devices.
Changes from baseline in biochemical parameters of oxidative stress and inflammation (at the end of ozone therapy). | At the end of ozone therapy (approx. week 16).
  Changes in serum levels of oxidative stress parameters (superoxide dismutase, glutathione, glutathione peroxidase, and free radicals) and proinflammatory cytokines.
Changes from baseline in biochemical parameters of oxidative stress and inflammation (at 12 weeks after the end of ozone therapy). | At 12 weeks after the end of ozone therapy (approx. week 28).
  Changes in serum levels of oxidative stress parameters (superoxide dismutase, glutathione, glutathione peroxidase, and free radicals) and proinflammatory cytokines.
Change from Baseline in Gut Microbiota Composition (at the end of ozone therapy). | At the end of ozone therapy (approx. week 16).
  Analysis of stool samples to evaluate changes in the intestinal microbiome (in patients treated with rectal ozone).
Change from Baseline in Gut Microbiota Composition (at 12 weeks after the end of ozone therapy). | At 12 weeks after the end of ozone therapy (approx. week 28).
  Analysis of stool samples to evaluate changes in the intestinal microbiome (in patients treated with rectal ozone).

CONTACTS AND LOCATIONS:
Overall Officials: Bernardino Clavo, MD, PhD, Study Chair — Dr. Negrín University Hospital, Las Palmas, Spain; Francisco Rodríguez-Esparragón, BSc, PhyD, Principal Investigator — Dr. Negrín University Hospital, Las Palmas, Spain; Ángeles Cánovas-Molina, RN, Principal Investigator — Dr. Negrín University Hospital, Las Palmas, Spain
Locations (1):
- Dr. Negrín University Hospital, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: Yes
* It will be available (after request): Individual participant data (IPD) that underlie the results reported in further articles, after deidentification
  * Data will be available after publication, ending 36 months following the article publication.
  * They will be available for investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available after publication, ending 36 months following article publication.
Access Criteria: They will be available for investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.

REFERENCES:
- [Result] Clavo B, Cordoba-Lanus E, Martinez-Sanchez G, Federico M, Canovas-Molina A, Pinero JE, Vargas-Prado AM, Ramchandani A, Zajac M, Ribeiro I, Navarro M, Jorge IJ, Gonzalez-Martin JM, Martin-Alfaro R, Fernandez-Tagarro M, Diaz-Garrido JA, Lorenzo-Morales J, Rodriguez-Esparragon F. Modulating the Gut Microbiota via Rectal Ozone Insufflation in Gynecological Cancer Patients with Radiotherapy/Chemotherapy-Induced Pelvic Toxicity: A Proposed Clinical Study Protocol. J Clin Med. 2025 Nov 12;14(22):8015. doi: 10.3390/jcm14228015. PMID 41303051
- [Result] Clavo B, Canovas-Molina A, Federico M, Martinez-Sanchez G, Benitez G, Galvan S, Ramallo-Farina Y, Fabelo H, Cazorla-Rivero S, Lago-Moreno E, Antonilli C, Diaz-Garrido JA, Jorge IJ, Marrero-Callico G, Rodriguez-Abreu D, Rodriguez-Esparragon F. Ozone Treatment in the Management of Chemotherapy-Induced Peripheral Neuropathy: A Review of Rationale and Research Directions. Cancers (Basel). 2025 Jul 8;17(14):2278. doi: 10.3390/cancers17142278. PMID 40723162
- [Result] Bisshopp S, Linertova R, Carames MA, Szolna A, Jorge IJ, Navarro M, Melchiorsen B, Rodriguez-Diaz B, Gonzalez-Martin JM, Clavo B. Pain Relief, Disability, and Hospital Costs After Intradiscal Ozone Treatment or Microdiscectomy for Lumbar Disc Herniation: A 24-Month Real-World Prospective Study. J Clin Med. 2025 Jun 26;14(13):4534. doi: 10.3390/jcm14134534. PMID 40648907
- [Result] Clavo B, Canovas-Molina A, Garcia-Lourve C, Cazorla-Rivero S, Federico M, Rodriguez-Esparragon F. Effects of ozone treatment on chemotherapy-induced peripheral neuropathy: a promising research area. Med Gas Res. 2025 Jun 1;15(2):195-197. doi: 10.4103/mgr.MEDGASRES-D-24-00074. Epub 2025 Jan 18. No abstract available. PMID 40070187
- [Result] Clavo B, Rodriguez-Abreu D, Galvan-Ruiz S, Federico M, Canovas-Molina A, Ramallo-Farina Y, Antonilli C, Benitez G, Fabelo H, Garcia-Lourve C, Gonzalez-Beltran D, Jorge IJ, Rodriguez-Esparragon F, Callico GM. Long-Term Effects of Ozone Treatment in Patients with Persistent Numbness and Tingling Secondary to Chemotherapy-Induced Peripheral Neuropathy. A Retrospective Study. Integr Cancer Ther. 2025 Jan-Dec;24:15347354241307038. doi: 10.1177/15347354241307038. PMID 39797612
- [Result] Clavo B, Canovas-Molina A, Diaz-Garrido JA, Canas S, Ramallo-Farina Y, Laffite H, Federico M, Rodriguez-Abreu D, Galvan S, Garcia-Lourve C, Gonzalez-Beltran D, Carames MA, Hernandez-Fleta JL, Serrano-Aguilar P, Rodriguez-Esparragon F. Effects of ozone therapy on anxiety and depression in patients with refractory symptoms of severe diseases: a pilot study. Front Psychol. 2023 Aug 4;14:1176204. doi: 10.3389/fpsyg.2023.1176204. eCollection 2023. PMID 37599784
- [Result] Clavo B, Rodriguez-Abreu D, Galvan S, Federico M, Martinez-Sanchez G, Ramallo-Farina Y, Antonelli C, Benitez G, Rey-Baltar D, Jorge IJ, Rodriguez-Esparragon F, Serrano-Aguilar P. Long-term improvement by ozone treatment in chronic pain secondary to chemotherapy-induced peripheral neuropathy: A preliminary report. Front Physiol. 2022 Aug 30;13:935269. doi: 10.3389/fphys.2022.935269. eCollection 2022. PMID 36111149
- [Result] Clavo B, Canovas-Molina A, Ramallo-Farina Y, Federico M, Rodriguez-Abreu D, Galvan S, Ribeiro I, Marques da Silva SC, Navarro M, Gonzalez-Beltran D, Diaz-Garrido JA, Cazorla-Rivero S, Rodriguez-Esparragon F, Serrano-Aguilar P. Effects of Ozone Treatment on Health-Related Quality of Life and Toxicity Induced by Radiotherapy and Chemotherapy in Symptomatic Cancer Survivors. Int J Environ Res Public Health. 2023 Jan 13;20(2):1479. doi: 10.3390/ijerph20021479. PMID 36674232
- [Result] Clavo B, Gutierrez D, Martin D, Suarez G, Hernandez MA, Robaina F. Intravesical ozone therapy for progressive radiation-induced hematuria. J Altern Complement Med. 2005 Jun;11(3):539-41. doi: 10.1089/acm.2005.11.539. PMID 15992242
- [Result] Clavo B, Suarez G, Aguilar Y, Gutierrez D, Ponce P, Cubero A, Robaina F, Carreras JL. Brain ischemia and hypometabolism treated by ozone therapy. Forsch Komplementmed. 2011;18(5):283-7. doi: 10.1159/000333795. Epub 2011 Oct 13. PMID 22105041
- [Result] Clavo B, Ceballos D, Gutierrez D, Rovira G, Suarez G, Lopez L, Pinar B, Cabezon A, Morales V, Oliva E, Fiuza D, Santana-Rodriguez N. Long-term control of refractory hemorrhagic radiation proctitis with ozone therapy. J Pain Symptom Manage. 2013 Jul;46(1):106-12. doi: 10.1016/j.jpainsymman.2012.06.017. Epub 2012 Oct 26. PMID 23102757
- [Result] Clavo B, Santana-Rodriguez N, Gutierrez D, Lopez JC, Suarez G, Lopez L, Robaina F, Bocci V. Long-term improvement in refractory headache following ozone therapy. J Altern Complement Med. 2013 May;19(5):453-8. doi: 10.1089/acm.2012.0273. Epub 2012 Dec 7. PMID 23215625
- [Result] Clavo B, Santana-Rodriguez N, Llontop P, Gutierrez D, Ceballos D, Mendez C, Rovira G, Suarez G, Rey-Baltar D, Garcia-Cabrera L, Martinez-Sanchez G, Fiuza D. Ozone Therapy in the Management of Persistent Radiation-Induced Rectal Bleeding in Prostate Cancer Patients. Evid Based Complement Alternat Med. 2015;2015:480369. doi: 10.1155/2015/480369. Epub 2015 Aug 18. PMID 26357522
- [Result] Clavo B, Santana-Rodriguez N, Llontop P, Gutierrez D, Suarez G, Lopez L, Rovira G, Martinez-Sanchez G, Gonzalez E, Jorge IJ, Perera C, Blanco J, Rodriguez-Esparragon F. Ozone Therapy as Adjuvant for Cancer Treatment: Is Further Research Warranted? Evid Based Complement Alternat Med. 2018 Sep 9;2018:7931849. doi: 10.1155/2018/7931849. eCollection 2018. PMID 30271455
- [Result] Clavo B, Rodriguez-Esparragon F, Rodriguez-Abreu D, Martinez-Sanchez G, Llontop P, Aguiar-Bujanda D, Fernandez-Perez L, Santana-Rodriguez N. Modulation of Oxidative Stress by Ozone Therapy in the Prevention and Treatment of Chemotherapy-Induced Toxicity: Review and Prospects. Antioxidants (Basel). 2019 Nov 26;8(12):588. doi: 10.3390/antiox8120588. PMID 31779159
- [Result] Clavo B, Navarro M, Federico M, Borrelli E, Jorge IJ, Ribeiro I, Rodriguez-Melcon JI, Carames MA, Santana-Rodriguez N, Rodriguez-Esparragon F. Ozone Therapy in Refractory Pelvic Pain Syndromes Secondary to Cancer Treatment: A New Approach Warranting Exploration. J Palliat Med. 2021 Jan;24(1):97-102. doi: 10.1089/jpm.2019.0597. Epub 2020 May 5. PMID 32379556
- [Result] Clavo B, Navarro M, Federico M, Borrelli E, Jorge IJ, Ribeiro I, Rodriguez-Melcon JI, Carames MA, Santana-Rodriguez N, Rodriguez-Esparragon F. Long-Term Results with Adjuvant Ozone Therapy in the Management of Chronic Pelvic Pain Secondary to Cancer Treatment. Pain Med. 2021 Sep 8;22(9):2138-2141. doi: 10.1093/pm/pnaa459. No abstract available. PMID 33738491
- [Result] Clavo B, Martinez-Sanchez G, Rodriguez-Esparragon F, Rodriguez-Abreu D, Galvan S, Aguiar-Bujanda D, Diaz-Garrido JA, Canas S, Torres-Mata LB, Fabelo H, Tellez T, Santana-Rodriguez N, Fernandez-Perez L, Marrero-Callico G. Modulation by Ozone Therapy of Oxidative Stress in Chemotherapy-Induced Peripheral Neuropathy: The Background for a Randomized Clinical Trial. Int J Mol Sci. 2021 Mar 10;22(6):2802. doi: 10.3390/ijms22062802. PMID 33802143